CLINICAL TRIAL: NCT02931266
Title: Evaluation of the Efficacy and Safety of the PASS MIS® System in the Treatment of Spinal Thoracolumbar Fractures
Brief Title: PASS MIS® Post-market Clinical Follow-up
Status: Terminated | Type: Observational
Why Stopped: Lack of inclusions
Sponsor: Medicrea International (Industry)
Responsible Party: Sponsor
Other Study IDs: 1102
Record Dates: First submitted 2016-06-27; First posted 2016-10-13 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Spinal Fractures
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PASS MIS® — Posterior mini-invasive osteosynthesis

SUMMARY:
Prospective, multicenter non comparative and observational study (post-market clinical follow-up).

DETAILED DESCRIPTION:
Patients operated with PASS MIS® manufactured by MEDICREA® INTERNATIONAL between July 2016 and July 2017.

The inclusion period will be 12 months and the follow-up 24 months

ELIGIBILITY:
Inclusion Criteria:

* Patient which need to be operated to treat a fracture at the lumbar and/or thoracic spine with the PASS MIS® device from MEDICREA®
* Patient > 18years
* Patient with a mature skeleton
* Patient able to understand the protocol and the planning visit
* Patient able to complete a self-administered questionnaire
* Patient who have signed the informed consent form

Exclusion Criteria:

* Patient presenting other medical indication than thoracolumbar fracture
* Patient unable or who refuse to sign an informed consent form
* Patient unable to complete a self-administered questionnaire
* Patient judged as non-compliant by the investigator or not able to come back for follow-up visits
* Patient who need to receive or who received an open procedure
* Patient who has been not implanted with the PASS MIS® system
* Pregnant women or intending to get pregnant within the next 2 years after the surgery
* Patient with contra-indications to do radiographies
* Local infectious state
* Allergy or intolerance to the materials, suspected or known
* Any contra-indications present in the notice of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suffering from thoraco-lumbar spinal fracture and receiving a posterior osteosynthesis through a mini-invasive approach
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Spinal stability | 12 months postoperatively
  To evaluate though X-rays, the efficacy of the device to promote the stability of the instrumented segments.
Spinal fusion | 12 months postoperatively
  Radiological assessment of bony fusion

SECONDARY OUTCOMES:
Adverse events | During surgery, 1-6 months, 12 months, 24 months postoperatively
  To quantify and describe adverse events
Disability | 1-6 months, 12 months, 24 months postoperatively
  To assess patients' disability through ODI questionnaire
Patient satisfaction index | 1-6 months, 12 months, 24 months postoperatively
  To assess patient satisfaction after surgery using a questionnaire
Pain | 1-6 months, 12 months, 24 months postoperatively
  To assess patient's pain using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Fuentes, MD, Principal Investigator — Hopital la Timone, Marseille
Locations (1):
- Hopital la Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: No